CLINICAL TRIAL: NCT01459276
Title: A Randomized, Active Controlled, Double-blind, Multi-Centre Study to Evaluate Safety and Immunogenicity of One Dose of FLUVAL AB-like (Trivalent, Whole Virus, Aluminium Phosphate Gel Adjuvanted) Influenza Vaccine Containing 6μgHA of Seasonal A/H1N1, A/H3N2 and B Influenza Antigens in Non-elderly Adult and Elderly Subjects
Brief Title: A Study to Evaluate Safety and Immunogenicity of FluvalAB-like Influenza Vaccine in Non-Elderly Adult and Elderly Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fluart Innovative Vaccine Ltd, Hungary (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: FluvalAB-H-15; 2011-003314-16 (EudraCT Number)
Record Dates: First submitted 2011-10-19; First posted 2011-10-25 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Influenza
Keywords: seasonal; prevention; influenza; infection; influenza vaccine; vaccine; influenza in humans
MeSH Terms: conditions — Influenza, Human; Infections | interventions — Vaccination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- FAB-6011 (Experimental): One 0.5 mL injection of FAB-6011 trivalent influenza vaccine containing 6μg HA of seasonal A/H1N1, A/H3N2 and B influenza antigens
  Interventions: Biological: Vaccination with FAB-6011
- FLUVALAB (Active Comparator): One 0.5 mL injection of FLUVAL AB trivalent influenza vaccine containing 15μg HA of seasonal A/H1N1, A/H3N2 and B influenza antigens
  Interventions: Biological: Vaccination with FluvalAB

INTERVENTIONS:
Biological: Vaccination with FAB-6011 — One 0.5 mL injection of FAB-6011 trivalent influenza vaccine containing 6μgHA of seasonal A/H1N1, A/H3N2 and B influenza antigens.
  Other Names: FAB-6011
  Arms: FAB-6011
Biological: Vaccination with FluvalAB — One 0.5 mL injection of FLUVAL AB trivalent influenza vaccine containing 15μgHA of seasonal A/H1N1, A/H3N2 and B influenza antigens.
  Other Names: FluvalAB
  Arms: FLUVALAB

SUMMARY:
The purpose of this study is to determine the immunogenicity and tolerability of one 0.5 mL intramuscular (IM) injection of FLUVAL AB-like trivalent influenza vaccine containing 6μgHA of seasonal A/H1N1, A/H3N2 and B influenza antigens in adults and elderly people.

ELIGIBILITY:
Inclusion Criteria:

* male and female adult volunteers aged 18 years or older,
* mentally competent,
* able to understand and comply with all study requirements,
* willing and able to give written informed consent prior to initiation of study procedures,
* in good health (as determined by clinical judgement of the investigator on the basis of medical history and existing medical condition) or are in stable medical condition. Subjects will not be excluded with known, adequately treated, clinically significant organ or systemic diseases (e.g. asthma or diabetes), such that, in the opinion of the investigator, the significance of the disease will not compromise the subject's participation in the study.
* Female subjects aged 18 to 60 years (i.e. participants of childbearing potential) with a negative result from the urine pregnancy test prior to vaccination who agrees to use an acceptable contraception method or abstinence throughout the trial and not become pregnant for the duration of the study.
* Absence of existence of any exclusion criteria.

Exclusion Criteria:

* Pregnancy, breast-feeding or positive urine pregnancy test at baseline prior to vaccination. Female subjects who are able to bear children but not willing to use an acceptable contraception method for the duration of the study.
* Hypersensitivity to eggs, chicken protein, thiomersal, formaldehyde, gentamycin, ciprofloxacin, neomycin or any other component of the vaccine;
* History of anaphylactic shock or neurological symptoms or signs following administration of any vaccine;
* History of Guillain-Barré syndrome;
* Serious disease, such as cancer, autoimmune disease, advanced arteriosclerotic disease, complicated diabetes mellitus, acute or progressive hepatic disease, acute or progressive renal disease, congestive heart failure;
* Immunosuppressive therapy within the past 36 months;
* Concomitant corticosteroid therapy, including high-dose inhaled corticosteroids;
* Receipt of immunostimulants;
* Receipt of parenteral immunoglobulin, blood products and/or plasma derivates within the past 3 months;
* Suspected or known HIV, HBV or HCV infection;
* Acute disease and/or axillary temperature ≥37oC within the past 3 days;
* Vaccine therapy within the past 4 weeks;
* Influenza vaccination (any kind) within the past 6 months;
* Experimental drug therapy within the past 4 weeks;
* Concomitant participation in another clinical study;
* Any condition which, in the opinion of the investigator, may interfere with the evaluation of the study;
* Past or current psychiatric disease of the subject that upon judgement of the investigator may have effect on the objective decision-making of the subject;
* Alcohol or drug abuse of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1206 (Actual)
Dates: Start 2011-10; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Measures of immunogenicity | 21-28 days following vaccination
  The measures of immunogenicity (by using HI test) are:
  * the GMTs at Day 0 and at Day 21
  * the Day 21/Day 0 geometric mean titer ratios (GMTRs)
  * the percentage of subjects achieving seroconversion or significant increase in antibody titer at Day 21
  * the percentage of subjects achieving a titer ≥40 at Day 0 and at Day 21.
Measures of safety | 21-28 days following vaccination
  The measures of safety are:
  Number and percentage of subjects with at least
  * one local reaction between Day 0 and Day 7
  * one systemic reaction between Day 0 and Day 7
  * one adverse event between Day 0 and visit at Day 21.

SECONDARY OUTCOMES:
Measures of long term immunogenicity | 110-120 days following vaccination
  The measures of long term immunogenicity (by using HI test) are:
  * the GMTs at Day 0 and at Day 120
  * the Day 120/Day 0 geometric mean titer ratios (GMTRs)
  * the percentage of subjects achieving seroconversion or significant increase in antibody titer at Day 120
  * the percentage of subjects achieving a titer ≥40 at Day 0 and at Day 120.
Measures of long term safety | 110-120 days following vaccination
  The measures of long term safety are:
  Number and percentage of subjects with at least
  * one local reaction
  * one systemic reaction
  * one adverse event between Day 0 and visit at Day 120.

CONTACTS AND LOCATIONS:
Overall Officials: Gabor Kollar, MD, Study Director — Omninvest Ltd; Ferenc Tamás, MD, Principal Investigator — Family Doctor's Office, Pilisvörösvár; Ágnes Hasitz, MD, Principal Investigator — Family Doctor's Office, Szentendre; Judit Simon, MD, Principal Investigator — Family Doctor's Office, Budapest; Barna Bőze, MD, Principal Investigator — Family Doctor's Office, Hatvan; Tibor Hrutka, MD, Principal Investigator — Family Doctor's Office, Vecsés; Péter Torzsa, MD, Principal Investigator — Family Doctor's Office, Budapest; Péter Vajer, MD, Principal Investigator — Family Doctor's Office, Biatorbágy
Locations (6):
- Hungary (6):
  - Péter Vajer, Biatorbágy, Pest County
  - Barna Bőze, Hatvan, Pest County
  - Family Doctor's Office, Szentendre, Pest County
  - Tibor Hrutka, Vecsés, Pest County
  - Family Doctor's Office, Budapest
  - Family Doctor's Office, Pilisvörösvár